CLINICAL TRIAL: NCT04443374
Title: The Reliability and Validity of the Turkish Version of the Simple Physical Activity Questionnaire (SIMPAQ)
Brief Title: The Turkish Version of the Simple Physical Activity Questionnaire (SIMPAQ)
Acronym: SIMPAQ
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Aybike Senel, PT,MSc, Research Assistant, Istanbul University - Cerrahpasa
Other Study IDs: 24
Record Dates: First submitted 2020-06-22; First posted 2020-06-23 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Psychiatric Disorder
Keywords: physical activity; measurement; assessment; sedentary behaviour; mental illness
MeSH Terms: conditions — Mental Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Simple Physical Activity Questionnaire (SIMPAQ) was originally developed in English to assess physical activity level particularly people with mental illnesses. The purpose of this study was to translate and cross-culturally adapt the SIMPAQ into Turkish and investigate its psychometric properties.

DETAILED DESCRIPTION:
The Simple Physical Activity Questionnaire (SIMPAQ) was originally developed in English to assess physical activity level particularly people with mental illnesses. The purpose of this study was to translate and cross-culturally adapt the SIMPAQ into Turkish and investigate its psychometric properties. Eighty individuals with mental illnesses (major depression, bipolar disorder, anxiety disorder, schizophrenia, alcohol and substance addiction) will include. For cross-cultural adaptation and validation procedure, developers' manual in the official site will be followed (http://www.simpaq.org/). Within a 5-to-7-day period after the first assessment, the participants completed the Turkish version of the SIMPAQ to evaluate test-retest reliability. Cronbach's alpha (α) was used to assess internal consistency. The correlations with the Turkish version of the International Physical Activity-Short Form (IPAQ-SF) and Brief Psychiatric Rating Scale (BPRS) and Turkish version of the DSM-5 Self-Rated Level 1 Cross-Cutting Symptom Scale-Adult Version (DSM XC) will determine to check the validity.

ELIGIBILITY:
Inclusion Criteria:

Aged between 18 and 60 years Being a volunteer to participate Being an outpatient or inpatient at the place of the study Being diagnosed with major depression, bipolar disorder, anxiety disorder, schizophrenia, alcohol and substance addiction according to DSM-5 or ICD.

Exclusion Criteria:

Having cognitive impairment Having disabilities in understanding, speaking and reading Turkish Having vision and / or hearing problems

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will include 80 patients diagnosed with major depression, bipolar disorder, anxiety disorder, schizophrenia, alcohol and substance addiction by the psychiatrists in Prof. Dr. Mazhar Osman Mental Health and Neurological Diseases Training and Research Hospital, University of Health Sciences. The individuals who volunteers and meets the inclusion criteria will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-08-02 (Actual)

PRIMARY OUTCOMES:
Simple Physical Activity Questionnaire | Baseline (First assessment)
  The SIMPAQ is a reliable and valid tool to assess physical activity in people with mental illness. The 5-item SIMPAQ was designed to capture activity over a representative 24-h period from the previous 7-days. Time spent in bed overnight, time sedentary, including napping, time spent walking, time spent exercising and time engaged in incidental activity are questioned and the sum of them should be approximately 24 h. This structure of the SIMPAQ provides interviewers to understand under or over-reporting. For an estimate of total self-reported moderate-vigorous physical activity (MVPA) time, time spent walking and exercising were combined to provide total MVPA (hours per week).

SECONDARY OUTCOMES:
Simple Physical Activity Questionnaire | Within a 5-to-7-day period after the first assessment (Second assessment)
  The SIMPAQ is a reliable and valid tool to assess physical activity in people with mental illness. The 5-item SIMPAQ was designed to capture activity over a representative 24-h period from the previous 7-days. Time spent in bed overnight, time sedentary, including napping, time spent walking, time spent exercising and time engaged in incidental activity are questioned and the sum of them should be approximately 24 h. This structure of the SIMPAQ provides interviewers to understand under or over-reporting. For an estimate of total self-reported moderate-vigorous physical activity (MVPA) time, time spent walking and exercising were combined to provide total MVPA (hours per week).
International Physical Activity Questionnaire-Short Form | Baseline (First assessment)
  International Physical Activity Questionnaire-Short Form (IPAQ-SF) is a self-report questionnaire that assesses PA in the last 7 days. IPAQ-SF provides information on walking, moderate and vigorous activities and time spent sitting, within a week.
Brief Psychiatric Rating Scale | Baseline (First assessment)
  Brief Psychiatric Rating Scale (BPRS) is a valid 18-item quantitative scale for assessing psychopathology and its severity. Each item is measured on a five-point scale (0 = none to 4 = very severe), with lower scores meaning a lower severity of the symptom.
DSM-5 Level 1 Cross-Cutting Symptom Measure-Adult | Baseline (First assessment)
  DSM-5 Level 1 Cross-Cutting Symptom Measure-Adult (DSM XC) comprises 23 self-rated symptoms that capture 13 mental health domains. Respondents indicate how much (or how often) they have been bothered by each symptom in the prior two weeks using a five-point response scale (none, not at all to severe, nearly every day). A score of 2 or higher in most domains, except substance use (score of 1 or higher) is suggestive of clinically-relevant mental health problems.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru KAYA MUTLU, PT, PhD, Study Director — İstanbul University-Cerrahpaşa
Locations (1):
- İstanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)